CLINICAL TRIAL: NCT00916539
Title: Non-displaced Scaphoid Fractures: A Clinical Trial of Cast Immobilization Including vs. Excluding the Thumb
Brief Title: Cast Immobilization for Non-Displaced Scaphoid Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006P-001424; IRB 2006p001424
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Non-displaced Scaphoid Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cast that immobilizes the thumb (Experimental): Cast that immobilizes the thumb
  Interventions: Device: Cast that immobilizes the thumb
- Cast that does not immobilize the thumb (Active Comparator): Cast that does not immobilize the thumb
  Interventions: Device: Cast that does not immobilize the thumb

INTERVENTIONS:
Device: Cast that immobilizes the thumb — Cast that immobilizes the thumb
  Arms: Cast that immobilizes the thumb
Device: Cast that does not immobilize the thumb — Cast that does not immobilize the thumb
  Arms: Cast that does not immobilize the thumb

SUMMARY:
This trial is trying to understand if immobilization of the thumb after a non-displaced scaphoid fracture affects recovery. The standard of care overseas is a cast that allows for free movement of the thumb, and in the United States it is a cast that immobilizes the thumb. This study is attempting to understand if there is a difference.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Isolated fracture of the scaphoid
3. No displacement of the scaphoid fracture on CT scan

Exclusion Criteria:

1. Associated ipsilateral ligament injury or fracture
2. Pregnant Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Ring, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusettes General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (14) | 42 (18) | 37.5 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 22 | 21 | 43
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Extent of Union
Description: The investigators looked at the extent of fracture union after immobilization.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: percentage of union
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
percentage of union | 70 (30) | 85 (24)

2. Secondary Outcome: DASH Questionnaire
Description: This questionnaire measures the disability of the upper extremity. The disability scale is ranked from 0 (least disability) to 100 (most disability).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
units on a scale | 5 (8) | 6 (9)

3. Secondary Outcome: Modified Mayo Wrist Score
Description: The Modified Mayo Wrist Score evaluates wrist function after treatment. The total score ranges from 0 to 100, with higher scores indicating a better result.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
units on a scale | 92 (9) | 87 (19)

4. Secondary Outcome: Grip Strength
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
kilograms | 40 (21) | 37 (21)

5. Secondary Outcome: Visual Analog Scale for Pain
Description: The pain scale measures the amount of pain on a scale from 0 to 10, where 10 indicates the most pain and 0 is no pain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
units on a scale | 1.1 (1.4) | 0.8 (1.3)

6. Secondary Outcome: Range of Motion: Flexion
Description: Range of motion measures the ability to move the wrist joint after injury.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
degrees | 76 (12) | 72 (9)

7. Secondary Outcome: Range of Motion: Extension
Description: Range of motion measures the ability to move the wrist joint after injury.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
degrees | 68 (15) | 67 (14)

8. Secondary Outcome: Range of Motion: Ulnar Deviation
Description: Range of motion measures the ability to move the wrist joint after injury.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
degrees | 38 (13) | 32 (8)

9. Secondary Outcome: Range of Motion: Radial Deviation
Description: Range of motion measures the ability to move the wrist joint after injury.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Number analyzed (Participants) | 31 | 31
degrees | 20 (9) | 19 (7)

ADVERSE EVENTS:
Arm/Group | Cast That Immobilizes the Thumb | Cast That Does Not Immobilize the Thumb
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No